CLINICAL TRIAL: NCT01395784
Title: Effects of Pioglitazone, a PPARgamma Receptor Agonist, on the Abuse Liability of Oxycodone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 6106; R01DA09236 (Other: NIH Grant Award Number)
Record Dates: First submitted 2011-07-13; First posted 2011-07-18 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2013-11

CONDITIONS: Opioid Abuse
Keywords: Oxycodone; Opioid abuse
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo Maintenance Period (Placebo Comparator): Participants will complete the various outcome measures following a 2-3 week maintenance period on Placebo (PCB).
  Interventions: Drug: pioglitazone
- PIO 15 Maintenance Period (Experimental): Participants will complete the various outcome measures following a 2-3 week maintenance period on Pioglitazone (PIO) 15 mg.
  Interventions: Drug: pioglitazone
- PIO 45 Maintenance Period (Experimental): Participants will complete the various outcome measures following a 2-3 week maintenance period on Pioglitazone (PIO) 45 mg.
  Interventions: Drug: pioglitazone

INTERVENTIONS:
Drug: pioglitazone — A PPARγ agonist, also marketed as Actos. Participants will be maintained on ascending doses of Placebo, pioglitazone 15 mg and 45 mg, prior to completing a lab session at the end of each dosing period.
  Other Names: Actos

SUMMARY:
The ability of pioglitazone (PIO) to alter the effects of opioids in humans has not been characterized in a controlled laboratory setting. Accordingly, the proposed investigation seeks to examine the effects of PIO on oxycodone, one of the most commonly used and abused opioid drugs in the U.S. (Davis et al., 2003). More specifically, the primary aim of this investigation is to characterize the subjective effects of oxycodone under maintenance on various doses of PIO (0, 15, and 45 mg) in non-dependent, prescription opioid abusers. Secondary aims of the study are to examine the influence of PIO on the analgesic, cognitive, and physiological effects of oxycodone.

DETAILED DESCRIPTION:
This 9-week investigation will use an inpatient/outpatient design in which participants will be maintained on ascending doses of pioglitazone (3 weeks on placebo followed by 3 weeks on PIO 15 mg followed by 3 weeks on PIO 45 mg). At the end of each maintenance period the effects of oxycodone (0, 10, and 20 mg) will be examined during a single laboratory session using a cumulative dosing procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Recreational use of prescription opioids at least once per month within the past year
2. No current major mood, psychotic, or anxiety disorder
3. Physically healthy
4. aspartate aminotransferase (AST) or alanine aminotransferase (ALT) within normal limits
5. Able to perform study procedures 6.21-45 years of age

7.Blood glucose concentration between 70-145 mg/dl for men and 70-125 mg/dl for women (fasting) 8.Hb > 13 for men and Hb > 11 for women with no other evidence of medical disorder resulting in blood loss or anemia/hematological disease

Exclusion Criteria:

1. Physical dependence on any drugs, excluding nicotine and caffeine
2. Participants requesting treatment
3. Participants on parole or probation
4. Pregnancy or lactation: Female participants must agree to the use of a barrier control method of contraception (e.g. male and female condoms, diaphragms, cervical caps and contraceptive sponges used in combination with spermicide)
5. Current or recent history of significant violent behavior (within the past 6 months)
6. Current major Axis I psychopathology that might interfere with ability to participate in the study
7. Significant suicide risk
8. Current chronic pain
9. Current or history of congestive heart failure, edema, or diabetes mellitus
10. Sensitivity, allergy, or contraindication to opioids or pioglitazone
11. Unstable physical disorders that might make participation hazardous, such as end-stage AIDS, hypertension (blood pressure > 140/90), or heart disease (please note that participants will be asked about previous visits to a cardiologist, chest pain, or strong palpitations; if these exist, they will be referred to a cardiologist and excluded unless cleared for participation by a cardiologist)

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-08; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D Comer, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia Univ/ NYSPI Division on Substance Abuse, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data has been presented at conferences and being prepared for a peer-review publication.

RESULTS

PARTICIPANT FLOW:
Groups:
- Withing-subjects, Placebo-Controlled: Participants will complete the various outcome measures following maintenance period of: Placebo, Pioglitazone 15 mg, and 45 mg.
  pioglitazone: A PPARγ agonist, also marketed as Actos.
Period: Overall Study
Arm/Group | Withing-subjects, Placebo-Controlled
Started | 32
Completed | 17
Not Completed | 15
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Population: Recreational prescription opioid users.
Groups:
- Withing-subjects, Placebo-Controlled: Participants will complete the various outcome measures following maintenance period of: Placebo, Pioglitazone 15 mg, and 45 mg.
Arm/Group | Withing-subjects, Placebo-Controlled
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Subjective Ratings of "Good" Drug Effect
Description: Visual analog scale ratings (0-100 mm scale, 0=Not at all, 100=Extremely)
Time Frame: Measured during the lab session conducted at the end of each maintenance period
Population: Shown below are peak drug effects from each of the 3 maintenance periods (Placebo, Pioglitazone (PIO) 15, and PIO 45)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Participants: Participants will complete the various outcome measures following maintenance period of: Placebo, Pioglitazone 15 mg, and 45 mg.
Arm/Group | All Participants
Number analyzed (Participants) | 17
units on a scale
  Placebo | 37 (12)
  PIO 15 | 35 (9)
  PIO 45 | 35 (11)

2. Secondary Outcome: Analgesic Responses Using the Cold Pressor Test
Description: Latency to withdraw hand from cold water during the cold pressor test.
Time Frame: Measured during the lab session conducted at the end of each maintenance period
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | All Participants
Number analyzed (Participants) | 17
seconds
  Placebo | 110 (23)
  PIO 15 | 71 (8)
  PIO 45 | 75 (10)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed daily throughout the study.
Description: A study nurse queried participants concerning any adverse events using the Systematic Assessment for Treatment Emergent Events (SAFTEE)
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No